CLINICAL TRIAL: NCT07030283
Title: Intraperitoneal Paclitaxel With Standard Systemic NALIRIFOX for Pancreatic Ductal Adenocarcinoma With Peritoneal Carcinomatosis: Prospective Pilot Trial
Brief Title: Intraperitoneal Paclitaxel With NALIRIFOX for Pancreatic Ductal Adenocarcinoma With Peritoneal Carcinomatosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-2111.cc
Record Dates: First submitted 2025-05-21; First posted 2025-06-22 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: Peritoneal Carcinomatosis; pancreatic adenocarcinoma; pancreatic ductal adenocarcinoma; PDAC; metastatic; NALIRIFOX; intraperitoneal chemotherapy; intraperitoneal paclitaxel; circulating tumor DNA (ctDNA); peritoneal cell-free DNA
MeSH Terms: conditions — Peritoneal Neoplasms; Neoplasm Metastasis | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intraperitoneal Paclitaxel with Systemic NALIRIFOX (Experimental): Intraperitoneal paclitaxel will be administered on days 1 and 8 via the intraperitoneal port, and systemic NALIRIFOX (Fluorouracil Continuous Infusion/Leucovorin/Liposomal Irinotecan/Oxaliplatin) will be administered on day 1 of each 14-day cycle. The maximum treatment duration is 12 cycles.
  Interventions: Drug: Paclitaxel; Drug: NALIRIFOX

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel is a chemotherapy medication that is FDA-approved to treat a number of cancer types. In this study, paclitaxel will be administered via the intraperitoneal port. Intraperitoneal paclitaxel is not FDA approved for pancreatic cancer.
  Other Names: Taxol
Drug: NALIRIFOX — NALIRIFOX is a systemic chemotherapy treatment for metastatic pancreatic cancer that was approved by the FDA in February 2024. It's a combination of drugs that are already approved to treat pancreatic cancer: Liposomal irinotecan (Nal-IRI or Onivyde®), 5 fluorouracil (5-FU)/leucovorin, and Oxaliplatin.

SUMMARY:
This goal of this clinical trial is to learn whether the drug combination of intraperitoneal paclitaxel (chemotherapy given directly into the abdominal cavity) and intravenous NALIRIFOX (chemotherapy given into a vein, including fluorouracil, leucovorin, oxaliplatin, and liposomal irinotecan) is safe and works in adults with pancreatic cancer that has spread to the peritoneum.

The main questions it aims to answer are:

* Are people with pancreatic cancer able to tolerate the combination drug regimen?
* How well does the combination drug regimen work to treat pancreatic cancer?

Participants will:

* Obtain a port that goes into the abdomen to deliver intraperitoneal paclitaxel (called an intraperitoneal catheter)
* Receive treatment with intravenous NALIRIFOX once every 2 weeks and intraperitoneal paclitaxel on days 1 and 8 of each 14-day cycle
* Visit the clinic with each treatment for checkups and laboratory testing
* Have imaging scans and blood lab testing to determine response to treatment
* Have abdominal fluid lab testing that may help determine if the cancer is responding to treatment
* Fill out questionnaires to see how the treatment affects how participants feel and function
* Continue follow up after treatment ends to track survival

Some participants may be able to have surgery later if the cancer responds well. This is called conversion surgery. To be eligible for surgery, the cancer must have shrunk or stayed the same, peritoneal fluid (from the abdomen) must no longer show cancer cells, and a tumor marker called CA 19-9 must decrease or return to normal. The decision to do surgery will depend on the treating surgeon.

By testing this new treatment strategy, researchers hope to find a safer and more effective way to treat people with pancreatic cancer that has spread to the abdomen. If successful, this approach may lead to longer survival, better quality of life, and more people becoming eligible for surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be age 18 years or older.
4. Histologically or cytologically confirmed pancreatic adenocarcinoma with histologically or cytologically proven seeding in the peritoneal cavity without metastasis to other organs.
5. Primary tumor that is resectable, borderline resectable, or locally advanced per NCCN classification.
6. PCI score ≤ 8.
7. ECOG performance status of 0 or 1
8. Prior treatment for 0-4 months with FOLFIRINOX, modified FOLFIRINOX, or NALIRIFOX and able to receive additional treatment per investigator opinion
9. Adequate biological parameters as evidenced by all of the following blood counts:

   * Absolute neutrophil count (ANC) >/= 1,500 per cubic millimeter without the use of hematopoietic growth factors within 14 days prior to screening
   * Platelet count >/= 75,000 per cubic millimeter
   * Hemoglobin > 9 g/dL
10. Adequate hepatic function as evidenced by:

    * Serum total bilirubin ≤ 1.5x ULN (biliary drainage is allowed for biliary obstruction), and
    * AST and ALT ≤ 3 x ULN
11. Adequate renal function as evidenced by serum creatinine <1.5 x ULN

Exclusion Criteria:

1. Prior treatment of pancreatic cancer in the metastatic setting with surgery or investigational therapy (Note: biliary drainage, diagnostic laparoscopy/laparotomy, and duodenal stenting is allowed).
2. Evident distant metastatic disease outside of the peritoneal cavity.
3. Extensive metastatic disease in peritoneal cavity (PCI>8).
4. Known disease progression with any prior chemotherapy.
5. Known hypersensitivity to paclitaxel or other liposomal products.
6. Current use of strong CYP2C8 inhibitors or inducers, or presence of any other contraindications for paclitaxel.
7. Known UGT1A1 deficiency or DPD deficiency.
8. Neuropathy Grade 2 or higher
9. Known active COVID infection with symptoms.
10. Has ever received or is currently receiving radiation for pancreatic cancer treatment.
11. Receipt of live, attenuated vaccine within 30 days prior the first dose of Intraperitoneal paclitaxel. (Note: enrolled patients should not receive live vaccines during the study and up to 30 days after the last dose of intraperitoneal paclitaxel).
12. Known positive test results for human immunodeficiency (HIV) or patients with chronic or active hepatitis B or C. Patients who have a history of hepatitis B or C who have undetectable HBV DNA or HCV RNA after anti-viral therapy may be enrolled.
13. Active infection during screening visits or on the day of treatment, which in the investigator's opinion might compromise the patient's participation in the trial or affect the study outcome.
14. Any other medical or social condition deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.
15. Pregnant or breast feeding; females of child-bearing potential must test negative for pregnancy within 7 days prior to C1D1. Both male and female patients of reproductive potential must agree to use a highly effective method of birth control during the study and for 9 months following the last dose of both IP PTX and IV NALIRIFOX.
16. Histologies other than adenocarcinoma, such as neuroendocrine (carcinoid, islet cell) or acinar pancreatic carcinoma.
17. Patients who, in the opinion of the investigator, have symptoms or signs suggestive of clinically unacceptable deterioration of the primary disease at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12-31 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2030-07-01 (Estimated)

PRIMARY OUTCOMES:
Adverse event rate | From enrollment through 30 days after last dose of treatment administered (approximately 7 months)

SECONDARY OUTCOMES:
1-year survival rate | From enrollment through 12 months after the last dose of treatment (approximately 18 months)
Overall survival | From enrollment through 24 months after the last dose of treatment (approximately 30 months)
Progression-free survival | From enrollment through end of treatment (approximately 6 months)
Objective response rate | From enrollment through end of treatment (approximately 6 months)
Change in peritoneal carcinomatosis index | From enrollment to 6 months after end of treatment (approximately 12 months)
  The peritoneal carcinomatosis index is a score used to assess the amount of cancer in the peritoneal cavity. The score ranges from 0 to 39, with a higher score indicating a greater extent of cancer.

OTHER OUTCOMES:
Changes in serum circulating tumor DNA | From enrollment to end of treatment (approximately 6 months)
Conversion surgery rate | From enrollment to end of treatment (approximately 6 months)
Change in quality of life assessed by EORTC QLQ-C30 questionnaire | From enrollment to 6 months after end of treatment (approximately 12 months)
  The EORTC QLQ-C30 is a validated questionnaire. Scores range from 0 (minimum) to 100 (maximum). Higher scores indicate worse symptoms on symptom scales and better functioning on functional scales.
Change in quality of life assessed by EORTC QLQ-PAN26 questionnaire | From enrollment to 6 months after end of treatment (approximately 12 months)
  The EORTC QLQ-PAN26 is a validated questionnaire. Scores range from 0 (minimum) to 100 (maximum). Higher scores indicate worse symptoms on symptom scales and better functioning on functional scales.
Changes in peritoneal cell-free DNA | From enrollment to end of treatment (approximately 6 months)
Changes in tumor markers (CEA and CA 19-9) | From enrollment to end of treatment (approximately 6 months)
Changes in peritoneal cytology | From enrollment to end of treatment (approximately 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Leal, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States